CLINICAL TRIAL: NCT01748305
Title: Moderate-to-vigorous Physical Activity for Glycemic Control in Patients With Gestational Diabetes Mellitus: a Pilot Study
Brief Title: Moderate-to-vigorous Physical Activity for Glycemic Control in Patients With Gestational Diabetes Mellitus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment issues.
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Antonio E. Frias, MD, MFM, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: e8631
Record Dates: First submitted 2012-12-10; First posted 2012-12-12 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Gestational Diabetes Mellitus; Exercise
Keywords: GDM; A1GDM; A2GDM
MeSH Terms: conditions — Diabetes, Gestational; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Moderate-to-vigorous intensity exercise (Experimental): Moderate-to-vigorous intensity exercise three times per day for three weeks
  Interventions: Behavioral: Moderate-to-vigorous intensity exercise

INTERVENTIONS:
Behavioral: Moderate-to-vigorous intensity exercise — Moderate-to-vigorous intensity exercise three times per day for three weeks

SUMMARY:
Patients with newly diagnosed gestational diabetes will be recruited. The control group with get routine diet and exercise counseling. The intervention group will be instructed to get moderate-to-vigorous intensity exercise; they will walk on a treadmill one time with supervision in order to be instructed how hard to work. All participants will keep an exercise log for 3 weeks and will wear an accelerometer for 1 week. The primary outcome is glucose control, specifically the need for medication in treatment of their diabetes. The hypothesis is that moderate or greater intensity exercise will better control glucose and lead to less need for medication management.

ELIGIBILITY:
Inclusion Criteria:

* gestational diabetes mellitus
* singelton pregnancy
* 18 years old or older
* no medical contraindications to exercise

Exclusion Criteria:

* multiple gestation
* non-English speaking
* unable to exercise
* preexisting diabetes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Need for medication for diabetes | 3 weeks

SECONDARY OUTCOMES:
Birth weight | delivery
A1c | delivery
Mode of delivery | delivery

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Frias, MD, Principal Investigator — Oregon Health and Science University; Jessica Voge, MD, Study Director — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States